CLINICAL TRIAL: NCT02513758
Title: Penetration and Compartimentation of HIV in Genital Mucosa
Brief Title: Penetration and Compartimentation of HIV
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 0201078; DGS 2002/0521 (Other: Health general direction)
Record Dates: First submitted 2015-07-30; First posted 2015-08-03 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: HIV
Keywords: HIV patients; Genital HIV penetration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood, saliva, sperm and cervicovaginal secretions
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HIV patients: Men will have blood sampling tubes of 10 ml each, a saliva sample and a sample of sperm Women will have a two blood sampling tubes of 10 ml each, a saliva sample and a sampling cervicovaginal secretions
  Interventions: Other: sample

INTERVENTIONS:
Other: sample — Men will have blood sampling tubes of 10 ml each, a saliva sample and a sample of sperm Women will have a two blood sampling tubes of 10 ml each, a saliva sample and a sampling cervicovaginal secretions

SUMMARY:
Genital mucosa is the main way of HIV penetration. Many cells can be involved (epithelial cells, Langerhans cells) and antibodies may also play a critical role. The investigators' study aims to precise the role of each type of cells, the interaction cell-cell and cell-antibodies.

DETAILED DESCRIPTION:
At inclusion, men will have a two blood sampling tubes of 10 ml each, a saliva sample and a sample of sperm and women will have a two blood sampling tubes of 10 ml each, a saliva sample and a sampling cervicovaginal secretions

ELIGIBILITY:
Inclusion Criteria:

* Adults (> 18 year-old) HIV positive,
* HIV-CV> 1000 cp/ml,

Exclusion Criteria:

* children

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV patients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2002-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Viral tropism of HIV | Inclusion
  number of HIV virus in sperm or cervical secretions.

SECONDARY OUTCOMES:
Genetic polymorphism for HIV strains | Inclusion
  With a sequencing method, it is possible to classify the different strains in groups, according to their polymorphism.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric LUCHT, PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- LUCHT, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No